CLINICAL TRIAL: NCT03670680
Title: Evaluation of the Efficiency of Lina LibrataTM System in the Treatment of Functional Idiopathic Menometrorrhagia
Brief Title: Efficiency of Lina LibrataTM System
Acronym: THERMOLIB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL17_0266; 2017-A02017-46 (Other: ID-RCB)
Record Dates: First submitted 2018-09-04; First posted 2018-09-13 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Menorrhagia
Keywords: Menorrhagia; Lina LibrataTM; efficiency; menometrorrhagia
MeSH Terms: conditions — Menorrhagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lina LibrataTM (Experimental): Use of the Lina LibrataTM
  Interventions: Device: Use of the Lina LibrataTM

INTERVENTIONS:
Device: Use of the Lina LibrataTM — Use of the Lina LibrataTM

SUMMARY:
Menometrorrhagia is the first cause of consultation in gynecology. Etiology of menometrorrhagia is varied, but in majority of cases no underlying pathology is found, they are said functional idiopathic menometrorrhagia .

In case of failure of medical treatment, for women who do not wish to preserve reproduction possibilities, a surgical treatment by endometrectomy (destruction of the uterine endometrial epithelial) can be proposed. Currently, a new system, Lina LibrataTM is available on the market. This system allows destructing endometrial membrane with a balloon which offer several advantages compared to present used system. Specially, it does not require dilatation of uterus's cervix and it reduces the pain. The investigator make hypothesis that the use of the system Lina LibrataTM does not cause pain and can be thus used under local anesthetic in ambulatory surgery. With the aim of developing ambulatory care, the main objective of this prospective monocentric study is to estimate the efficiency of Lina LibrataTM system in the treatment of functional idiopathic menometrorrhagia. Secondary objectives are to estimate the pain during the procedure, the rate of per and post-complications and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Women from 40 to 50 years old
* Not menopausal women
* Do not want pregnancy
* Having dysfunctional bleeding
* informed and signed consent

Exclusion Criteria:

* Unacceptable postoperative risk disclosed on interview: coagulation disorder, immune disorder, evolutive disease, etc
* Pregnancy or wish to have later pregnancy
* Endometrium cancer (or suspicious of cancer) or precancerous conditions of the endometrium
* Anatomical conditions (i-e history of caesarian, transmural myomectomy) or pathological conditions (i-e long term treatment) which can weaken myometrium
* Genital or urinary infection at the time of the procedure
* Intra uterine device
* Pelvic inflammation
* Inability to understand information provided
* Not covered by a national health insurance scheme, prisoner or under administrative supervision

Ages: 38 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
rate of amenorrhea | 4 weeks

SECONDARY OUTCOMES:
pain score | during surgery (Hour 0)
  Pain at Hour 0 is assessed by VAS (Visual Analog Scale) rating from 0 to 10 (0=no pain).
pain score | 2 hours after surgery (Hour 2)
  Pain at Hour 2 is assessed by VAS (Visual Analog Scale) rating from 0 to 10 (0=no pain).
pain score | 6 hours after surgery (Hour 6)
  Pain at Hour 6 is assessed by QDSA (Questionnaire de la Douleur Saint-Antoine).
pain score | 6 hours after surgery (Hour 6)
  Pain at Hour 6 1 is assessed by VAS (Visual Analog Scale) rating from 0 to 10 (0=no pain)..
pain score | the day after surgery (Day 1)
  Pain at Day 1 is assessed by QDSA (Questionnaire de la Douleur Saint-Antoine).
pain score | the day after surgery (Day 1)
  Pain at Day 1 is assessed by VAS (Visual Analog Scale) rating from 0 to 10 (0=no pain).
pain score | one week after surgery (Day 7)
  Pain at Day 7 is assessed by QDSA (Questionnaire de la Douleur Saint-Antoine)
pain score | one week after surgery (Day 7)
  Pain at Day 7 is assessed by VAS (Visual Analog Scale) rating from 0 to 10 (0=no pain).
pain score | one month after surgery (Month 1)
  Pain at Month 1 is assessed by QDSA (Questionnaire de la Douleur Saint-Antoine)
pain score | one month after surgery (Month 1)
  Pain at Month 1 is assessed by VAS (Visual Analog Scale) rating from 0 to 10 (0=no pain).
recurrences of menorrhagia | at month 1
recurrences of menorrhagia | at month 6
assessment of menorrhagia on Higham's score | 1 month after surgery
  Assessment by patients on Higham's score. A score greater than 100 points corresponds to bleeding greater than 80 ml of blood.
assessment of menorrhagia on Higham's score | 6 months after surgery
  Assessment by patients on Higham's score. A score greater than 100 points corresponds to bleeding greater than 80 ml of blood.
evolution of hemoglobinemia | 1 month after surgery
  hemoglobin measured by blood test
evolution of hemoglobinemia | 6 months after surgery
  hemoglobin measured by blood test
per-operative complications | per surgery day 0
post-operative complications | post surgery day 0
measure of quality of life | at month 1
  assessed by the questionnaire SF-12 (abridged version of the Medical Outcomes Study Short-Form General Health Survey SF-36). It allows to obtain 2 scores: mental and social score (from 5.89058 to 71.966825) and physical score (from 9.94738 to 70.02246). The average of this scores in the general population is 50.
measure of quality of life | at month 6
  assessed by the questionnaire SF-12 (abridged version of the Medical Outcomes Study Short-Form General Health Survey SF-36). It allows to obtain 2 scores: mental and social score (from 5.89058 to 71.966825) and physical score (from 9.94738 to 70.02246). The average of this scores in the general population is 50.
measure of symptoms improvement | at month 1
  assessed by the questionnaire PGI-I (from 1 "much better" to 7 "much worse")
measure of symptoms improvement | at month 6
  assessed by the questionnaire PGI-I (from 1 "much better" to 7 "much worse")

CONTACTS AND LOCATIONS:
Overall Officials: Géry LAMBLIN, MD, Principal Investigator — Hospices Civils de Lyon Gynaecology Department
Locations (1):
- Hospices Civils de Lyon, Bron, France